CLINICAL TRIAL: NCT05518565
Title: Exploration of the Length/Tension Relationship in Spastic Muscle in Vivo and Its Relation to the Muscle's Macromolecular Composition. The Results Are Related to Function Before and After Tendon Transfer/Tendon Lengthenings.
Brief Title: The Muscle in Cerebral Palsy; Sarcomere Length in Vivo and Microscopic Characterization of Biopsies.
Acronym: CPMuscleSL
Status: Recruiting | Type: Observational
Sponsor: Eva Ponten (Other Government)
Responsible Party: Sponsor-Investigator, Eva Ponten, MD PhD Ass Prof, Region Stockholm
Organization: Region Stockholm (Other Government)
Other Study IDs: CP muskel OP laser
Record Dates: First submitted 2022-07-27; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Cerebral Palsy; Muscle Contracture; Spasticity, Muscle
Keywords: Cerebral Palsy; Muscle biopsy; Laser diffraction; Sarcomere Length; Muscle contracture
MeSH Terms: conditions — Cerebral Palsy; Contracture; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Muscle biopsies taken during surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Cerebral palsy (CP) is a motor impairment due to a brain malformation or a brain lesion before the age of two. Spasticity, hypertonus in flexor muscles, dyscoordination and an impaired sensorimotor control are cardinal symptoms. The brain lesion is non-progressive, but the flexor muscles of the limbs will during adolescence become relatively shorter and shorter (contracted), forcing the joints into a progressively flexed position. This will worsen the positions of already paretic and malfunctioning arms and legs. Due to bending forces across the joints, bony malformations will occur, worsening the function even further. Currently, the initial treatment of choice is the use of braces, which diminishes the shortening somewhat, but eventually lengthenings of tendons and release of aponeuroses around the muscles often is needed, and transfers of wrist flexors to wrist extensors may improve wrist position. But the long-term results are unpredictable- how much does the muscle need to be lengthened? What muscles should be transferred for a better position of the wrist, and at what tension? A method to measure sarcomere length in vivo has been developed. The sarcomere, the distance between two striations, is the smallest contractile unit in the striated muscle. When, during surgery, a muscle fiber bundle is transilluminated with a low energy laser light, a diffraction pattern is formed. This diffraction pattern reflects the sarcomere length, and thereby an instant measure of how the stretch of the muscle is obtained. When performing tendon transfers of e.g. wrist flexors to wrist extensors, the setting of the tension of the transfer is arbitrary, and the long-term result is unpredictable. Laser diffraction measurements will give a guide to a precise setting of tension. It is known that there may be pathological changes in muscle in cerebral palsy that also will affect the long-term results of tendon lengthenings and transfers. In order to also take these changes into account, small muscle biopsies will be taken during the same surgeries. These will be examined with immuno-histochemical and biochemical techniques, gel-electrophoresis as well as electron microscopy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a motor impairment due to a brain malformation or a brain lesion before the age of two. Spasticity, hypertonus in flexor muscles, dyscoordination and an impaired sensorimotor control are cardinal symptoms. The brain lesion is non-progressive, but the flexor muscles of the limbs will during adolescence become relatively shorter and shorter (contracted), forcing the joints into a progressively flexed position. This will worsen the positions of already paretic and malfunctioning arms and legs. Due to bending forces across the joints, bony malformations will occur, worsening the function even further. Currently, the initial treatment of choice is the use of braces, which diminishes the shortening somewhat, but eventually lengthenings of tendons and release of aponeuroses around the muscles often is needed, and transfers of wrist flexors to wrist extensors may improve wrist position. But the long-term results are unpredictable- how much does the muscle need to be lengthened? What muscles should be transferred for a better position of the wrist, and at what tension? A method to measure sarcomere length in vivo has been developed. The sarcomere, the distance between two striations, is the smallest contractile unit in the striated muscle. When, during surgery, a muscle fiber bundle is transilluminated with a low energy laser light, a diffraction pattern is formed. This diffraction pattern reflects the sarcomere length, and thereby an instant measure of how the stretch of the muscle is obtained. When performing tendon transfers of e.g. wrist flexors to wrist extensors, the setting of the tension of the transfer is arbitrary, and the long-term result is unpredictable. Laser diffraction measurements will give a guide to a precise setting of tension. It is known that there may be pathological changes in muscle in cerebral palsy that also will affect the long-term results of tendon lengthenings and transfers. In order to also take these changes into account, small muscle biopsies will be taken during the same surgeries. These will be examined with immuno-histochemical and biochemical techniques, gel-electrophoresis as well as electron microscopy.

Research questions:

* Is the muscle in CP different from muscle from typically developed children regarding architecture, protein expression and sarcomere length?
* Is there a difference between extensors and flexors?
* Are the contractile proteins (myosins) more altered in children with more severe CP, with a negative impact on endurance?
* Is growth potential negatively affected?
* Are the muscle fibers short and stretched out, contributing to poor muscle force?
* Is an increased amount of collagen in the muscle contributing to stiffness and changes in sarcomere length? The most important measurements: Sarcomere length in vivo, muscle fiber area, histochemical morphometry, muscle fiber types (immunohistochemistry), quantification of myosins with SDH gel electrophoresis, satellite cell detection, qRT-PCR and Western blotting to exploring gene expression.
* During surgeries that are planned according to clinical routines, muscles are that are necessary to expose in order to perform the surgery are investigated. Laser diffraction measurements are performed through the range of motion of adjacent joints. Muscle specimens 3x3 mm are taken at least 1 cm away from where the laser diffraction device (Myometer) was used.
* The muscle specimens are snap frozen and stored at -80°C until analyzed. The expression of different myosin heavy chain (MyHC) isoforms is assessed by using the monoclonal antibodies (mAb) N2.261, mAb A4.840 against slow MyHC I, mAb F1.652 against embryonic MyHC, and mAb NCL-MHCn against fetal (=neonatal) MyHC)(Tiger, Champliaud et al. 1997; Wewer, Thornell et al. 1997). Satellite cells will be identified with mAb against N-CAM (neural cell adhesion molecule). The fibers are typed according to the content of MyHCs.

Significance: Children with cerebral palsy have a motor impairment and progressive contractures that we often treat late; when tendon and bony surgery are the only options to realign the joints. More information on the muscle architecture, composition and growth potential will give more knowledge the reasons for increasing flexion contractures in children with cerebral palsy. With this knowledge, hopefully new treatment regimens and improved surgical techniques for this patient group can be developed.

ELIGIBILITY:
Inclusion Criteria:

* Celebral Palsy or Aquired Brain Injury

Exclusion Criteria:

* Progressive neurological disease

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children who due to clinical indications need surgery of the arm or the lower leg. Patients are consecutively recruited.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2002-01-15 (Actual); Primary Completion 2032-12-15 (Estimated); Study Completion 2033-12-15 (Estimated)

PRIMARY OUTCOMES:
Sarcomere lenght measurements intraooperatively in vivo with laser diffraction | One hour
  micrometer
Muscle biopsy structure, fiber area | one hour
  square mm
Muscle biopsy gene expression and protein content | one hour
  percentage %

CONTACTS AND LOCATIONS:
Overall Officials: Eva M Pontén, MD PhD, Principal Investigator — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Karolinska University Hospital, Stockholm
  - Karolinska University Hospitla, Stockholm
  - Karolinska, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided